CLINICAL TRIAL: NCT03547167
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by Administration of PNEUMOVAX™23 Six Months Later in Immunocompetent Adults Between 18 and 49 Years of Age at Increased Risk for Pneumococcal Disease (PNEU - DAY)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by PNEUMOVAX™23 in Adults at Increased Risk for Pneumococcal Disease (V114-017/PNEU-DAY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-017; 2017-004915-38 (EudraCT Number); V114-017 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2)
  Interventions: Biological: V114; Biological: PNEUMOVAX™23
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2)
  Interventions: Biological: Prevnar 13™; Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and Merck Aluminum Phosphate Adjuvant (125 mcg) in each 0.5 mL dose
  Arms: V114
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg), and aluminum phosphate adjuvant (125 mcg aluminum) in each 0.5 ml dose
  Other Names: PCV13
  Arms: Prevnar 13™
Biological: PNEUMOVAX™23 — 23-valent pneumococcal polysaccharide vaccine with serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F (25 mcg each) in each 0.5 mL dose
  Other Names: PPV23

SUMMARY:
This study is designed to 1) describe the safety, tolerability, and immunogenicity of V114 and Prevnar 13™ in pneumococcal vaccine-naïve adults at increased risk for pneumococcal disease and to 2) describe the safety, tolerability, and immunogenicity of PNEUMOVAX™23 when administered 6 months after receipt of either V114 or Prevnar 13™. Increased risk for pneumococcal disease is defined as 1) an underlying medical condition, 2) behavioral habits such as smoking or alcohol use, or 3) living in a community/environment with increased risk of disease transmission.

ELIGIBILITY:
Inclusion Criteria:

* Native American participant enrolled from any of the clinical sites of the Johns Hopkins Center for American Indian Health (CAIH) without any of the pre-specified risk conditions for pneumococcal disease listed below, OR Native American participant enrolled from any of the CAIH sites or participant from a site other than CAIH with ≥1 of the following risk conditions for pneumococcal disease:

  1. Diabetes mellitus Type 1 or Type 2 and with hemoglobin A1c (HgA1c) <10%
  2. Chronic liver disease with documented history of compensated cirrhosis (Child-Pugh Score A)
  3. Confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD) with spirometric Global Initiative for Chronic Obstructive Lung Disease Stage 1 to 3
  4. Confirmed diagnosis of mild or moderate persistent asthma receiving guideline directed therapy
  5. Confirmed diagnosis of chronic heart disease (New York Heart Association [NYHA] heart failure Class 1 to 3, receiving guideline-directed oral heart failure treatment) due to reduced or preserved ejection fraction or due to non-cyanotic congenital heart disease.
  6. Current smoker
* Female participant: not pregnant, not breastfeeding and 1) not of childbearing potential, or 2) of childbearing potential and agrees to practice contraception through 6 weeks after last administration of study vaccine.

Exclusion Criteria:

* History of active hepatitis within the prior 3 months
* History of diabetic ketoacidosis, or >1 episodes of severe, symptomatic hypoglycemia within the prior 3 months
* Myocardial infarction, acute coronary syndrome, transient ischemic attack, and ischemic or hemorrhagic stroke within the prior 3 months
* History of severe pulmonary hypertension or history of Eisenmenger syndrome
* History of invasive pneumococcal disease (IPD) or known history of other culture-positive pneumococcal disease within the prior 3 years
* Known hypersensitivity to any vaccine component, pneumococcal conjugate vaccine, or diphtheria toxoid-containing vaccine
* Known or suspected impairment of immunological function (including human immunodeficiency virus (HIV) infection or autoimmune disease)
* History of malignancy within the prior 5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* History of Stage 4 or 5 Chronic Kidney Disease or nephrotic syndrome
* History of alcohol withdrawal or alcohol withdrawal seizure within the prior 12 months
* History of coagulation disorder contraindicating intramuscular vaccination
* History of hospitalization within the prior 3 months
* Planned organ transplantation (heart, liver, lung, kidney, or pancreas) or other planned major surgery during the duration of this study.
* Expected survival for less than 1 year according to the investigator's judgment.
* Female participant: positive urine or serum pregnancy test
* Prior administration of any pneumococcal vaccine
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed within the prior 30 days
* Received systemic corticosteroids exceeding physiologic replacement doses within 14 days before study vaccination
* Receiving immunosuppressive or immunomodulatory therapy with a biological agent
* Received any licensed, non-live vaccine within 14 days before receipt of study vaccine or is scheduled to receive any licensed, non-live vaccine within 30 days following receipt of study vaccine
* Received any live vaccine within 30 days before receipt of any study vaccine or is scheduled to receive any live vaccine within 30 days following receipt of any study vaccine
* Received a blood transfusion or blood products within the prior 6 months
* Receiving chronic home oxygen therapy
* Participated in another clinical study of an investigational product within the prior 2 months
* Current user of recreational or illicit drugs or history of drug abuse or dependence
* Diabetes mellitus with HgA1c ≥10%
* Chronic liver disease with Child-Pugh Class B or C cirrhosis
* Chronic lung disease with Chronic Obstructive Pulmonary Disease (COPD) GOLD Stage 4 or severe persistent asthma
* Chronic heart disease with NYHA heart failure Class 4.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1515 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (78):
- United States (38):
  - Chinle Comprehensive Health Care Facility ( Site 0001), Chinle, Arizona
  - Fort Defiance Center for American Indian Health ( Site 0002), Fort Defiance, Arizona
  - Pulmonary Associates, PA ( Site 0043), Glendale, Arizona
  - Central Phoenix Medical Clinic, LLC ( Site 0031), Phoenix, Arizona
  - Whiteriver Center for American Indian Health ( Site 0005), Whiteriver, Arizona
  - Inland Empire Clinical Trials, LLC ( Site 0052), Rialto, California
  - Top Medical Research, Inc ( Site 0033), Cutler Bay, Florida
  - Indago Research & Health Center, Inc ( Site 0054), Hialeah, Florida
  - Renstar Medical Research ( Site 0008), Ocala, Florida
  - Triple O Research Institute, P.A. ( Site 0026), West Palm Beach, Florida
  - Emory University School of Medicine at Grady Hospital ( Site 0027), Atlanta, Georgia
  - Kootenai Health ( Site 0042), Coeur d'Alene, Idaho
  - Evanston Premier Healthcare & Research, LLC. ( Site 0012), Evanston, Illinois
  - Pharmakon Inc ( Site 0049), Evergreen Park, Illinois
  - Reid Physician Associates ( Site 0055), Richmond, Indiana
  - The Center for Pharmaceutical Research PC ( Site 0050), Kansas City, Missouri
  - Clinical Research Consortium ( Site 0053), Las Vegas, Nevada
  - Internal Medicine Associates [Bridgeton, NJ] ( Site 0015), Bridgeton, New Jersey
  - Gallup Center for American Indian Health ( Site 0003), Gallup, New Mexico
  - Shiprock Center for American Indian Health ( Site 0004), Shiprock, New Mexico
  - Corning Center For Clinical Research ( Site 0036), Corning, New York
  - Mid Hudson Medical Research ( Site 0022), New Windsor, New York
  - Wake Research Associates, LLC ( Site 0016), Raleigh, North Carolina
  - Lehigh Valley Health Network ( Site 0040), Allentown, Pennsylvania
  - University of Pennsylvania ( Site 0030), Philadelphia, Pennsylvania
  - Mountain View Clinical Research ( Site 0007), Greer, South Carolina
  - Holston Medical Group ( Site 0025), Kingsport, Tennessee
  - AIM Trials ( Site 0060), Fort Worth, Texas
  - University of Texas Medical Branch at Galveston ( Site 0034), Galveston, Texas
  - Private Practice Leadership, LLC ( Site 0051), Houston, Texas
  - Texas Center For Drug Development ( Site 0041), Houston, Texas
  - Texas Institute Of Cardiology ( Site 0048), McKinney, Texas
  - Village Health Partners ( Site 0006), Plano, Texas
  - Copperview Medical Center ( Site 0038), South Jordan, Utah
  - Timber Lane Allergy & Asthma Research, LLC ( Site 0044), South Burlington, Vermont
  - Pulmonary & Sleep Research ( Site 0046), Spokane Valley, Washington
  - Gundersen Health System ( Site 0021), La Crosse, Wisconsin
  - Marshfield Clinic ( Site 0013), Marshfield, Wisconsin
- Australia (6):
  - Paratus Clinical Pty Ltd - Blacktown Clinic ( Site 0174), Blacktown, New South Wales
  - Holdsworth House Medical Practice ( Site 0170), Sydney, New South Wales
  - Core Research Group Pty limited ( Site 0175), Brisbane, Queensland
  - Emeritus Research Pty Ltd ( Site 0173), Camberwell, Victoria
  - Paratus Clinical Kanwal ( Site 0172), Kanwal
  - Nepean Hospital ( Site 0176), Kingswood
- Canada (9):
  - The Liver and Intestinal Research Centre (LAIR) ( Site 0302), Vancouver, British Columbia
  - GA Research Associates, Ltd/Ltee ( Site 0303), Moncton, New Brunswick
  - Colchester Research Group ( Site 0094), Truro, Nova Scotia
  - Hamilton Medical Research Group ( Site 0092), Hamilton, Ontario
  - SKDS Research Inc. ( Site 0099), Newmarket, Ontario
  - Omnispec Recherche Clinique Inc ( Site 0093), Mirabel, Quebec
  - Dynamik Research ( Site 0095), Pointe-Claire, Quebec
  - Diex Recherche Quebec Inc ( Site 0091), Québec, Quebec
  - Q & T Research Sherbrooke Inc. ( Site 0097), Sherbrooke, Quebec
- Chile (5):
  - Clinica Arauco Salud ( Site 0100), Santiago, RM
  - Centro de Investigacion Clinica UC CICUC ( Site 0104), Santiago
  - CECIM ( Site 0101), Santiago
  - CESFAM Esmeralda ( Site 0102), Santiago
  - Hospital Dr. Hernan Henriquez Aravena ( Site 0105), Temuco
- New Zealand (8):
  - Southern Clinical Trials - Waitemata ( Site 0183), Auckland
  - Auckland Clinical Studies Limited ( Site 0189), Auckland
  - Optimal Clinical Trials ( Site 0182), Auckland
  - Christchurch Heart Institute ( Site 0280), Christchurch
  - Southern Clinical Trials Ltd ( Site 0180), Christchurch
  - Lakeland Clinical Trials ( Site 0181), Rotorua
  - Bay of Plenty Clinical School ( Site 0186), Tauranga
  - P3 Research Ltd - Wellington ( Site 0184), Wellington
- Poland (9):
  - WSOZ im.T.Browicza w Bydgoszczy ( Site 0317), Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz ( Site 0139), Bydgoszcz
  - Synexus Polska Sp. z o.o. ( Site 0238), Gdansk
  - Specjalistyczny osrodek .All-Med. Grazyna Pulka ( Site 0233), Krakow
  - ID Clinic ( Site 0235), Mysłowice
  - Centrum Medyczne Ogrodowa Sp. Z o.o. ( Site 0319), Skierniewice
  - Niepubliczny Zaklad Opieki Zdrowotnej ( Site 0314), Sopot
  - Wroclawskie Centrum Zdrowia SP ZOZ ( Site 0236), Wroclaw
  - Synexus Polska Sp. z o.o. oddział we Wrocławiu ( Site 0234), Wroclaw
- Russia (3):
  - Republican Clinical Hospital of Infectious Diseases n. a. A.F.Agafonov ( Site 0249), Kazan'
  - Saratov State Medical University n.a. V.I.Razumovskiy ( Site 0144), Saratov
  - Smolensk State Medical University ( Site 0246), Smolensk

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Hammitt LL, Quinn D, Janczewska E, Pasquel FJ, Tytus R, Rajender Reddy K, Abarca K, Khaertynova IM, Dagan R, McCauley J, Cheon K, Pedley A, Sterling T, Tamms G, Musey L, Buchwald UK. Immunogenicity, Safety, and Tolerability of V114, a 15-Valent Pneumococcal Conjugate Vaccine, in Immunocompetent Adults Aged 18-49 Years With or Without Risk Factors for Pneumococcal Disease: A Randomized Phase 3 Trial (PNEU-DAY). Open Forum Infect Dis. 2021 Dec 18;9(3):ofab605. doi: 10.1093/ofid/ofab605. eCollection 2022 Mar. PMID 35146039

RESULTS

PARTICIPANT FLOW:
Groups:
- V114: Participants were to receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
- Prevnar 13™: Participants were to receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 1135 | 380
Vaccination 1 - (V114 or Prevnar 13™, Day 1) | 1133 | 379
Vaccination 2 - (PNEUMOVAX™23, Month 6) | 1035 | 346
Completed | 1038 | 350
Not Completed | 97 | 30
Not completed — Withdrawal by Subject | 34 | 12
Not completed — Screen Failure | 0 | 1
Not completed — Lost to Follow-up | 59 | 15
Not completed — Death | 4 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 1135 | 380 | 1515
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.9) | 35.8 (8.9) | 35.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 581 | 201 | 782
  Male | 554 | 179 | 733
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 39 | 174
  Not Hispanic or Latino | 984 | 338 | 1322
  Unknown or Not Reported | 16 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 445 | 148 | 593
  Asian | 15 | 8 | 23
  Native Hawaiian or Other Pacific Islander | 33 | 11 | 44
  Black or African American | 43 | 18 | 61
  White | 582 | 192 | 774
  More than one race | 17 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events Following V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 1 with either V114 or Prevnar 13™, the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain. Estimated confidence intervals (CIs) are calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 5 days after Vaccination 1
Population: The analysis population included all randomized participants who received the relevant study vaccination for the timepoint of interest and were included in the intervention group according to the intervention they received. One participant in the Prevnar 13™ group incorrectly received V114 and was included in the V114 group for safety analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and were to receive a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and were to receive a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1134 | 378
Percentage of Participants
  Injection site redness/erythema | 15.1 [13.0 to 17.3] | 14.0 [10.7 to 17.9]
  Injection site tenderness/pain | 75.8 [73.2 to 78.3] | 68.8 [63.8 to 73.4]
  Injection site swelling | 21.7 [19.3 to 24.2] | 22.2 [18.1 to 26.8]

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following vaccination with V114 or Prevnar 13™, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. Estimated CIs are calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 14 days after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1134 | 378
Percentage of Participants
  Joint pain/arthralgia | 12.7 [10.8 to 14.8] | 11.6 [8.6 to 15.3]
  Tiredness/fatigue | 34.3 [31.5 to 37.1] | 36.8 [31.9 to 41.9]
  Headache | 26.5 [23.9 to 29.1] | 24.9 [20.6 to 29.5]
  Muscle pain/myalgia | 28.8 [26.2 to 31.6] | 25.5 [22.1 to 31.2]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Following V114 or Prevnar 13™
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator. Following vaccination with V114 or Prevnar 13™, the percentage of serious adverse events of V114 compared with Prevnar 13™ was assessed. Estimated CIs are calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to Month 6 (before Vaccination 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1134 | 378
Percentage of Participants | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.8]

4. Primary Outcome: Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity Day 30 Following V114 or Prevnar 13™
Description: The geometric mean titer (GMT) of serotype-specific opsonophagocytic activity (OPA) for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a multiplex opsonophagocytic assay. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Day 30
Population: The analysis population included all randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and had sufficient data to perform the analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 1019 | 341
  Serotype 1 (Shared) | 268.6 [243.7 to 296.0] | 267.2 [220.4 to 323.9]
  Serotype 3 (Shared): number analyzed (Participants) | 1004 | 340
  Serotype 3 (Shared) | 199.3 [184.6 to 215.2] | 150.6 [130.6 to 173.8]
  Serotype 4 (Shared): number analyzed (Participants) | 1016 | 342
  Serotype 4 (Shared) | 1416.0 [1308.9 to 1531.8] | 2576.1 [2278.0 to 2913.2]
  Serotype 5 (Shared): number analyzed (Participants) | 1018 | 343
  Serotype 5 (Shared) | 564.8 [512.7 to 622.2] | 731.1 [613.6 to 871.0]
  Serotype 6A (Shared): number analyzed (Participants) | 1006 | 335
  Serotype 6A (Shared) | 12928.8 [11923.4 to 14019.0] | 11282.4 [9718.8 to 13097.5]
  Serotype 6B (Shared): number analyzed (Participants) | 1014 | 342
  Serotype 6B (Shared) | 10336.9 [9649.4 to 11073.4] | 6995.7 [6024.7 to 8123.2]
  Serotype 7F (Shared): number analyzed (Participants) | 1019 | 342
  Serotype 7F (Shared) | 5756.4 [5410.4 to 6124.6] | 7588.9 [6775.3 to 8500.2]
  Serotype 9V (Shared): number analyzed (Participants) | 1015 | 343
  Serotype 9V (Shared) | 3355.1 [3135.4 to 3590.1] | 3983.7 [3557.8 to 4460.7]
  Serotype 14 (Shared): number analyzed (Participants) | 1016 | 343
  Serotype 14 (Shared) | 5228.9 [4847.6 to 5640.2] | 5889.8 [5218.2 to 6647.8]
  Serotype 18C (Shared): number analyzed (Participants) | 1014 | 343
  Serotype 18C (Shared) | 5709.0 [5331.1 to 6113.6] | 3063.2 [2699.8 to 3475.5]
  Serotype 19A (Shared): number analyzed (Participants) | 1015 | 343
  Serotype 19A (Shared) | 5369.9 [5017.7 to 5746.8] | 5888.0 [5228.2 to 6631.0]
  Serotype 19F (Shared): number analyzed (Participants) | 1018 | 343
  Serotype 19F (Shared) | 3266.3 [3064.4 to 3481.4] | 3272.7 [2948.2 to 3632.9]
  Serotype 23F (Shared): number analyzed (Participants) | 1016 | 340
  Serotype 23F (Shared) | 4853.5 [4469.8 to 5270.2] | 3887.3 [3335.8 to 4530.0]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 1005 | 320
  Serotype 22F (Unique to V114) | 3926.5 [3645.9 to 4228.7] | 291.6 [221.8 to 383.6]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 1014 | 338
  Serotype 33F (Unique to V114) | 11627.8 [10824.6 to 12490.7] | 2180.6 [1828.7 to 2600.2]

5. Secondary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events Following PNEUMOVAX™23
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following Vaccination 2 with PNEUMOVAX™23, the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain. Estimated CIs are calculated based on the exact binomial method proposed by Clopper and Pearson and are provided in accordance with the statistical analysis plan.
Time Frame: Up to 5 days after Vaccination 2 (Month 6)
Population: All randomized participants who received the relevant study vaccination for the timepoint of interest and were included in the intervention group according to the intervention they received. One participant in the Prevnar 13™ group incorrectly received V114 and was included in the V114 group for safety analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1036 | 345
Percentage of Participants
  Injection site redness/erythema | 22.6 [20.1 to 25.3] | 25.5 [21.0 to 30.5]
  Injection site tenderness/pain | 68.8 [65.9 to 71.6] | 67.0 [61.7 to 71.9]
  Injection site swelling | 29.4 [26.7 to 32.3] | 32.2 [27.3 to 37.4]

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events Following PNEUMOVAX™23
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Following Vaccination 2 with PNEUMOVAX™23, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue. Estimated CIs are calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 14 days after Vaccination 2 (Month 6)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1036 | 345
Percentage of Participants
  Joint pain/arthralgia | 12.0 [10.1 to 14.1] | 11.0 [7.9 to 14.8]
  Tiredness/fatigue | 30.1 [27.3 to 33.0] | 30.7 [25.9 to 35.9]
  Headache | 21.2 [18.8 to 23.9] | 21.2 [17.0 to 25.9]
  Muscle pain/myalgia | 24.1 [21.6 to 26.9] | 25.5 [21.0 to 30.5]

7. Secondary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Following PNEUMOVAX™23
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator. Following vaccination with PNEUMOVAX™23, the percentage of serious adverse events of V114 compared with Prevnar 13™ was assessed. Estimated CIs are calculated based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: From Month 6 (before Vaccination 2) to Month 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1036 | 345
Percentage of Participants | 0.0 [0.0 to 0.3] | 0.3 [0.0 to 1.6]

8. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Immunoglobulin G at Day 30
Description: The geometric mean concentration (GMC) of serotype-specific immunoglobulin G (IgG) for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 1 (Shared) | 3.56 [3.29 to 3.85] | 4.59 [4.00 to 5.26]
  Serotype 3 (Shared): number analyzed (Participants) | 1017 | 343
  Serotype 3 (Shared) | 0.77 [0.72 to 0.83] | 0.63 [0.57 to 0.71]
  Serotype 4 (Shared): number analyzed (Participants) | 1015 | 343
  Serotype 4 (Shared) | 1.53 [1.40 to 1.66] | 2.71 [2.34 to 3.13]
  Serotype 5 (Shared): number analyzed (Participants) | 1020 | 342
  Serotype 5 (Shared) | 3.43 [3.14 to 3.75] | 4.48 [3.77 to 5.32]
  Serotype 6A (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 6A (Shared) | 11.84 [10.71 to 13.10] | 10.87 [9.06 to 13.05]
  Serotype 6B (Shared): number analyzed (Participants) | 1020 | 342
  Serotype 6B (Shared) | 17.90 [16.21 to 19.76] | 11.36 [9.45 to 13.66]
  Serotype 7F (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 7F (Shared) | 5.18 [4.77 to 5.62] | 6.88 [5.95 to 7.95]
  Serotype 9V (Shared): number analyzed (Participants) | 1019 | 343
  Serotype 9V (Shared) | 4.44 [4.11 to 4.80] | 5.31 [4.62 to 6.10]
  Serotype 14 (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 14 (Shared) | 15.91 [14.46 to 17.51] | 17.35 [14.93 to 20.16]
  Serotype 18C (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 18C (Shared) | 14.57 [13.42 to 15.81] | 9.32 [8.06 to 10.79]
  Serotype 19A (Shared): number analyzed (Participants) | 1020 | 343
  Serotype 19A (Shared) | 19.41 [18.00 to 20.93] | 21.79 [18.85 to 25.19]
  Serotype 19F (Shared): number analyzed (Participants) | 1018 | 343
  Serotype 19F (Shared) | 13.98 [12.90 to 15.14] | 13.35 [11.52 to 15.47]
  Serotype 23F (Shared): number analyzed (Participants) | 1019 | 343
  Serotype 23F (Shared) | 13.57 [12.44 to 14.80] | 10.98 [9.34 to 12.91]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 1020 | 342
  Serotype 22F (Unique to V114) | 6.22 [5.74 to 6.74] | 0.52 [0.45 to 0.60]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 1020 | 342
  Serotype 33F (Unique to V114) | 7.79 [7.16 to 8.48] | 0.88 [0.78 to 1.00]

9. Secondary Outcome: Geometric Mean Fold Rise in Serotype-specific OPA Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a Multiplex Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 1001 | 334
  Serotype 1 (Shared) | 22.8 [20.6 to 25.1] | 21.9 [18.4 to 26.2]
  Serotype 3 (Shared): number analyzed (Participants) | 982 | 329
  Serotype 3 (Shared) | 5.8 [5.4 to 6.3] | 4.8 [4.3 to 5.5]
  Serotype 4 (Shared): number analyzed (Participants) | 988 | 329
  Serotype 4 (Shared) | 17.9 [16.2 to 19.8] | 33.4 [28.1 to 39.7]
  Serotype 5 (Shared): number analyzed (Participants) | 1003 | 337
  Serotype 5 (Shared) | 17.3 [15.7 to 18.9] | 21.1 [18.0 to 24.7]
  Serotype 6A (Shared): number analyzed (Participants) | 910 | 298
  Serotype 6A (Shared) | 21.7 [19.6 to 23.9] | 21.4 [18.0 to 25.5]
  Serotype 6B (Shared): number analyzed (Participants) | 969 | 328
  Serotype 6B (Shared) | 32.2 [28.6 to 36.3] | 25.0 [20.6 to 30.5]
  Serotype 7F (Shared): number analyzed (Participants) | 945 | 318
  Serotype 7F (Shared) | 7.3 [6.6 to 8.2] | 10.0 [8.3 to 12.0]
  Serotype 9V (Shared): number analyzed (Participants) | 977 | 332
  Serotype 9V (Shared) | 4.9 [4.5 to 5.3] | 5.7 [5.0 to 6.6]
  Serotype 14 (Shared): number analyzed (Participants) | 973 | 331
  Serotype 14 (Shared) | 8.2 [7.4 to 9.2] | 8.7 [7.2 to 10.6]
  Serotype 18C (Shared): number analyzed (Participants) | 973 | 331
  Serotype 18C (Shared) | 20.4 [18.6 to 22.4] | 11.7 [10.1 to 13.6]
  Serotype 19A (Shared): number analyzed (Participants) | 975 | 326
  Serotype 19A (Shared) | 12.5 [11.3 to 13.9] | 13.6 [11.4 to 16.2]
  Serotype 19F (Shared): number analyzed (Participants) | 985 | 329
  Serotype 19F (Shared) | 7.5 [6.9 to 8.2] | 7.4 [6.4 to 8.6]
  Serotype 23F (Shared): number analyzed (Participants) | 945 | 310
  Serotype 23F (Shared) | 22.5 [20.0 to 25.4] | 17.8 [14.6 to 21.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 885 | 290
  Serotype 22F (Unique to V114) | 13.9 [11.8 to 16.3] | 1.3 [1.1 to 1.6]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 979 | 326
  Serotype 33F (Unique to V114) | 5.4 [4.9 to 5.9] | 1.0 [0.8 to 1.1]

10. Secondary Outcome: GMFR in Serotype-specific IgG Day 1 to Day 30
Description: IgG for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 1 (Shared) | 12.2 [11.3 to 13.2] | 15.7 [13.9 to 17.8]
  Serotype 3 (Shared): number analyzed (Participants) | 1004 | 338
  Serotype 3 (Shared) | 4.1 [3.8 to 4.3] | 3.6 [3.2 to 4.0]
  Serotype 4 (Shared): number analyzed (Participants) | 1001 | 338
  Serotype 4 (Shared) | 8.0 [7.4 to 8.6] | 16.2 [14.3 to 18.4]
  Serotype 5 (Shared): number analyzed (Participants) | 1007 | 337
  Serotype 5 (Shared) | 4.3 [4.0 to 4.7] | 5.2 [4.5 to 6.0]
  Serotype 6A (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 6A (Shared) | 35.5 [32.5 to 38.8] | 31.3 [26.7 to 36.6]
  Serotype 6B (Shared): number analyzed (Participants) | 1006 | 337
  Serotype 6B (Shared) | 40.5 [37.1 to 44.2] | 28.0 [24.2 to 32.4]
  Serotype 7F (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 7F (Shared) | 12.2 [11.3 to 13.2] | 16.9 [14.8 to 19.3]
  Serotype 9V (Shared): number analyzed (Participants) | 1006 | 338
  Serotype 9V (Shared) | 10.6 [9.8 to 11.4] | 12.8 [11.3 to 14.5]
  Serotype 14 (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 14 (Shared) | 11.3 [10.3 to 12.5] | 11.5 [9.7 to 13.7]
  Serotype 18C (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 18C (Shared) | 30.5 [28.0 to 33.1] | 20.0 [17.2 to 23.2]
  Serotype 19A (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 19A (Shared) | 11.1 [10.2 to 12.0] | 14.0 [12.2 to 16.0]
  Serotype 19F (Shared): number analyzed (Participants) | 1005 | 338
  Serotype 19F (Shared) | 14.4 [13.2 to 15.7] | 15.3 [13.1 to 17.7]
  Serotype 23F (Shared): number analyzed (Participants) | 1006 | 338
  Serotype 23F (Shared) | 26.5 [24.2 to 29.0] | 22.0 [19.0 to 25.5]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 1007 | 337
  Serotype 22F (Unique to V114) | 11.4 [10.4 to 12.6] | 1.0 [1.0 to 1.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 1007 | 337
  Serotype 33F (Unique to V114) | 8.3 [7.7 to 8.9] | 1.0 [1.0 to 1.0]

11. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Day 1 to Day 30
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a Multiplexed Opsonophagocytic Assay. The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 1001 | 334
  Serotype 1 (Shared) | 83.9 [81.5 to 86.1] | 81.4 [76.8 to 85.5]
  Serotype 3 (Shared): number analyzed (Participants) | 982 | 329
  Serotype 3 (Shared) | 62.2 [59.1 to 65.3] | 56.8 [51.3 to 62.3]
  Serotype 4 (Shared): number analyzed (Participants) | 988 | 329
  Serotype 4 (Shared) | 79.0 [76.4 to 81.5] | 87.8 [83.8 to 91.2]
  Serotype 5 (Shared): number analyzed (Participants) | 1003 | 337
  Serotype 5 (Shared) | 83.4 [81.0 to 85.7] | 84.9 [80.6 to 88.5]
  Serotype 6A (Shared): number analyzed (Participants) | 910 | 298
  Serotype 6A (Shared) | 87.5 [85.1 to 89.6] | 85.2 [80.7 to 89.1]
  Serotype 6B (Shared): number analyzed (Participants) | 969 | 328
  Serotype 6B (Shared) | 84.7 [82.3 to 86.9] | 83.8 [79.4 to 87.7]
  Serotype 7F (Shared): number analyzed (Participants) | 945 | 318
  Serotype 7F (Shared) | 56.8 [53.6 to 60.0] | 64.5 [58.9 to 69.7]
  Serotype 9V (Shared): number analyzed (Participants) | 977 | 332
  Serotype 9V (Shared) | 51.5 [48.3 to 54.7] | 55.4 [49.0 to 60.8]
  Serotype 14 (Shared): number analyzed (Participants) | 973 | 331
  Serotype 14 (Shared) | 59.8 [56.7 to 62.9] | 60.4 [54.9 to 65.7]
  Serotype 18C (Shared): number analyzed (Participants) | 973 | 331
  Serotype 18C (Shared) | 84.5 [82.1 to 86.7] | 75.8 [70.8 to 80.3]
  Serotype 19A (Shared): number analyzed (Participants) | 975 | 326
  Serotype 19A (Shared) | 72.1 [69.2 to 74.9] | 75.2 [70.1 to 79.8]
  Serotype 19F (Shared): number analyzed (Participants) | 985 | 329
  Serotype 19F (Shared) | 64.3 [61.2 to 67.3] | 65.7 [60.2 to 70.8]
  Serotype 23F (Shared): number analyzed (Participants) | 945 | 310
  Serotype 23F (Shared) | 78.7 [76.0 to 81.3] | 77.7 [72.7 to 82.2]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 885 | 290
  Serotype 22F (Unique to V114) | 58.9 [55.5 to 62.1] | 15.5 [11.5 to 20.2]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 979 | 326
  Serotype 33F (Unique to V114) | 52.9 [49.7 to 56.1] | 3.1 [1.5 to 5.6]

12. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Day 1 to Day 30
Description: IgG for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. The percentage of participants who had ≥ 4-fold rise in IgG concentration are calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 1 (Shared) | 81.2 [78.7 to 83.6] | 86.4 [82.3 to 89.9]
  Serotype 3 (Shared): number analyzed (Participants) | 1004 | 338
  Serotype 3 (Shared) | 44.8 [41.7 to 48.0] | 41.1 [35.8 to 46.6]
  Serotype 4 (Shared): number analyzed (Participants) | 1001 | 338
  Serotype 4 (Shared) | 70.1 [67.2 to 73.0] | 86.1 [81.9 to 89.6]
  Serotype 5 (Shared): number analyzed (Participants) | 1007 | 337
  Serotype 5 (Shared) | 44.1 [41.0 to 47.2] | 50.4 [45.0 to 55.9]
  Serotype 6A (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 6A (Shared) | 93.3 [91.6 to 94.8] | 88.2 [84.2 to 91.4]
  Serotype 6B (Shared): number analyzed (Participants) | 1006 | 337
  Serotype 6B (Shared) | 93.4 [91.7 to 94.9] | 90.5 [86.9 to 93.4]
  Serotype 7F (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 7F (Shared) | 79.3 [76.7 to 81.8] | 86.4 [82.3 to 89.9]
  Serotype 9V (Shared): number analyzed (Participants) | 1006 | 338
  Serotype 9V (Shared) | 76.5 [73.8 to 79.1] | 84.0 [79.7 to 87.8]
  Serotype 14 (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 14 (Shared) | 70.8 [67.9 to 73.6] | 68.6 [63.4 to 73.6]
  Serotype 18C (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 18C (Shared) | 91.1 [89.1 to 92.8] | 87.3 [83.2 to 90.6]
  Serotype 19A (Shared): number analyzed (Participants) | 1007 | 338
  Serotype 19A (Shared) | 75.3 [72.5 to 77.9] | 82.0 [77.4 to 85.9]
  Serotype 19F (Shared): number analyzed (Participants) | 1005 | 338
  Serotype 19F (Shared) | 80.0 [77.4 to 82.4] | 80.8 [76.2 to 84.8]
  Serotype 23F (Shared): number analyzed (Participants) | 1006 | 338
  Serotype 23F (Shared) | 89.2 [87.1 to 91.0] | 87.6 [83.6 to 90.9]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 1007 | 337
  Serotype 22F (Unique to V114) | 73.1 [70.2 to 75.8] | 1.5 [0.5 to 3.4]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 1007 | 337
  Serotype 33F (Unique to V114) | 70.0 [67.1 to 72.8] | 0.3 [0.0 to 1.6]

13. Secondary Outcome: Geometric Mean Titer of Serotype-specific OPA at Month 7
Description: The geometric mean titer (GMT) of serotype-specific OPA for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a multiplex opsonophagocytic assay. The within-group 95% CIs are obtained by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 841 | 281
  Serotype 1 (Shared) | 266.6 [243.6 to 291.8] | 214.4 [180.7 to 254.5]
  Serotype 3 (Shared): number analyzed (Participants) | 837 | 279
  Serotype 3 (Shared) | 211.0 [195.2 to 228.1] | 208.0 [179.7 to 240.7]
  Serotype 4 (Shared): number analyzed (Participants) | 840 | 283
  Serotype 4 (Shared) | 1734.5 [1620.7 to 1856.4] | 1980.6 [1771.3 to 2214.6]
  Serotype 5 (Shared): number analyzed (Participants) | 844 | 283
  Serotype 5 (Shared) | 595.1 [544.5 to 650.5] | 626.7 [531.7 to 738.7]
  Serotype 6A (Shared): number analyzed (Participants) | 830 | 276
  Serotype 6A (Shared) | 5810.3 [5366.9 to 6290.3] | 5739.9 [4974.4 to 6623.1]
  Serotype 6B (Shared): number analyzed (Participants) | 843 | 283
  Serotype 6B (Shared) | 5215.2 [4863.6 to 5592.2] | 4412.4 [3892.8 to 5001.5]
  Serotype 7F (Shared): number analyzed (Participants) | 843 | 283
  Serotype 7F (Shared) | 6070.5 [5699.7 to 6465.6] | 6223.9 [5595.3 to 6923.0]
  Serotype 9V (Shared): number analyzed (Participants) | 842 | 282
  Serotype 9V (Shared) | 3133.1 [2918.4 to 3363.7] | 3364.1 [2972.2 to 3807.6]
  Serotype 14 (Shared): number analyzed (Participants) | 843 | 283
  Serotype 14 (Shared) | 5644.9 [5262.5 to 6055.2] | 5317.6 [4686.1 to 6034.1]
  Serotype 18C (Shared): number analyzed (Participants) | 842 | 281
  Serotype 18C (Shared) | 3260.6 [3057.3 to 3477.5] | 2294.4 [2052.5 to 2564.8]
  Serotype 19A (Shared): number analyzed (Participants) | 836 | 283
  Serotype 19A (Shared) | 4336.2 [4038.6 to 4655.6] | 4286.4 [3838.6 to 4786.4]
  Serotype 19F (Shared): number analyzed (Participants) | 844 | 282
  Serotype 19F (Shared) | 3198.6 [3011.0 to 3397.8] | 3085.4 [2770.7 to 3435.9]
  Serotype 23F (Shared): number analyzed (Participants) | 839 | 283
  Serotype 23F (Shared) | 3057.3 [2823.0 to 3311.0] | 2896.0 [2494.1 to 3362.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 837 | 280
  Serotype 22F (Unique to V114) | 3624.0 [3384.5 to 3880.3] | 4060.2 [3358.6 to 4908.4]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 837 | 282
  Serotype 33F (Unique to V114) | 11356.6 [10492.4 to 12291.9] | 16053.2 [13688.1 to 18827.1]

14. Secondary Outcome: Geometric Mean Concentration of Serotype-specific IgG at Month 7
Description: The geometric mean concentration (GMC) of serotype-specific immunoglobulin G (IgG) for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay.
Time Frame: Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 844 | 283
  Serotype 1 (Shared) | 2.91 [2.71 to 3.12] | 3.42 [3.02 to 3.87]
  Serotype 3 (Shared): number analyzed (Participants) | 844 | 283
  Serotype 3 (Shared) | 0.66 [0.62 to 0.71] | 0.68 [0.61 to 0.76]
  Serotype 4 (Shared): number analyzed (Participants) | 843 | 281
  Serotype 4 (Shared) | 1.33 [1.23 to 1.44] | 1.77 [1.55 to 2.02]
  Serotype 5 (Shared): number analyzed (Participants) | 844 | 283
  Serotype 5 (Shared) | 3.45 [3.17 to 3.75] | 3.92 [3.37 to 4.56]
  Serotype 6A (Shared): number analyzed (Participants) | 843 | 283
  Serotype 6A (Shared) | 4.25 [3.84 to 4.69] | 4.88 [4.08 to 5.85]
  Serotype 6B (Shared): number analyzed (Participants) | 844 | 283
  Serotype 6B (Shared) | 6.79 [6.15 to 7.49] | 6.04 [5.08 to 7.19]
  Serotype 7F (Shared): number analyzed (Participants) | 844 | 283
  Serotype 7F (Shared) | 3.46 [3.36 to 3.94] | 4.07 [3.54 to 4.68]
  Serotype 9V (Shared): number analyzed (Participants) | 844 | 283
  Serotype 9V (Shared) | 3.18 [2.96 to 3.43] | 3.61 [3.17 to 4.12]
  Serotype 14 (Shared): number analyzed (Participants) | 844 | 283
  Serotype 14 (Shared) | 14.28 [13.13 to 15.53] | 14.59 [12.64 to 16.85]
  Serotype 18C (Shared): number analyzed (Participants) | 844 | 283
  Serotype 18C (Shared) | 5.50 [5.07 to 5.98] | 4.24 [3.71 to 4.84]
  Serotype 19A (Shared): number analyzed (Participants) | 844 | 283
  Serotype 19A (Shared) | 11.26 [10.47 to 12.11] | 12.04 [10.57 to 13.72]
  Serotype 19F (Shared): number analyzed (Participants) | 844 | 283
  Serotype 19F (Shared) | 9.07 [8.45 to 9.74] | 8.81 [7.74 to 10.02]
  Serotype 23F (Shared): number analyzed (Participants) | 844 | 282
  Serotype 23F (Shared) | 5.42 [4.98 to 5.89] | 4.96 [4.25 to 5.81]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 844 | 283
  Serotype 22F (Unique to V114) | 4.85 [4.50 to 5.23] | 4.76 [4.01 to 5.65]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 844 | 283
  Serotype 33F (Unique to V114) | 5.98 [5.50 to 6.50] | 8.66 [7.31 to 10.26]

15. Secondary Outcome: GMFR in Serotype-specific OPA Day 1 to Month 7
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a Multiplexed Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 826 | 276
  Serotype 1 (Shared) | 22.6 [20.6 to 24.8] | 17.4 [14.8 to 20.5]
  Serotype 3 (Shared): number analyzed (Participants) | 820 | 270
  Serotype 3 (Shared) | 6.1 [5.6 to 6.6] | 6.4 [5.6 to 7.3]
  Serotype 4 (Shared): number analyzed (Participants) | 820 | 273
  Serotype 4 (Shared) | 21.6 [19.5 to 23.9] | 25.6 [21.7 to 30.3]
  Serotype 5 (Shared): number analyzed (Participants) | 831 | 279
  Serotype 5 (Shared) | 17.8 [16.3 to 19.3] | 18.3 [15.8 to 21.1]
  Serotype 6A (Shared): number analyzed (Participants) | 754 | 247
  Serotype 6A (Shared) | 9.6 [8.7 to 10.5] | 11.0 [9.3 to 13.0]
  Serotype 6B (Shared): number analyzed (Participants) | 802 | 273
  Serotype 6B (Shared) | 16.6 [14.7 to 18.7] | 15.7 [12.8 to 19.2]
  Serotype 7F (Shared): number analyzed (Participants) | 777 | 264
  Serotype 7F (Shared) | 7.7 [6.9 to 8.6] | 8.2 [6.7 to 9.9]
  Serotype 9V (Shared): number analyzed (Participants) | 810 | 273
  Serotype 9V (Shared) | 4.5 [4.2 to 4.9] | 4.9 [4.2 to 5.7]
  Serotype 14 (Shared): number analyzed (Participants) | 809 | 275
  Serotype 14 (Shared) | 9.2 [8.2 to 10.3] | 8.0 [6.6 to 9.7]
  Serotype 18C (Shared): number analyzed (Participants) | 805 | 273
  Serotype 18C (Shared) | 11.1 [10.2 to 12.2] | 9.1 [7.9 to 10.5]
  Serotype 19A (Shared): number analyzed (Participants) | 806 | 271
  Serotype 19A (Shared) | 9.6 [8.6 to 10.6] | 9.7 [8.1 to 11.6]
  Serotype 19F (Shared): number analyzed (Participants) | 818 | 272
  Serotype 19F (Shared) | 6.9 [6.3 to 7.6] | 7.1 [6.1 to 8.3]
  Serotype 23F (Shared): number analyzed (Participants) | 780 | 260
  Serotype 23F (Shared) | 14.0 [12.4 to 15.7] | 12.6 [10.3 to 15.4]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 742 | 254
  Serotype 22F (Unique to V114) | 12.1 [10.4 to 14.3] | 16.6 [12.2 to 22.6]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 810 | 273
  Serotype 33F (Unique to V114) | 5.1 [4.6 to 5.7] | 6.6 [5.5 to 8.0]

16. Secondary Outcome: GMFR in Serotype-specific IgG Day 1 to Month 7
Description: as for outcome 10
Time Frame: Day 1 (Baseline) and Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 1 (Shared) | 10.1 [9.4 to 10.8] | 11.4 [10.1 to 12.8]
  Serotype 3 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 3 (Shared) | 3.5 [3.3 to 3.7] | 3.8 [3.4 to 4.2]
  Serotype 4 (Shared): number analyzed (Participants) | 830 | 278
  Serotype 4 (Shared) | 7.1 [6.7 to 7.6] | 10.7 [9.5 to 12.0]
  Serotype 5 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 5 (Shared) | 4.3 [4.0 to 4.6] | 4.6 [4.1 to 5.2]
  Serotype 6A (Shared): number analyzed (Participants) | 832 | 280
  Serotype 6A (Shared) | 12.3 [11.3 to 13.4] | 13.9 [12.0 to 16.1]
  Serotype 6B (Shared): number analyzed (Participants) | 832 | 280
  Serotype 6B (Shared) | 15.3 [14.1 to 16.6] | 14.9 [13.0 to 17.0]
  Serotype 7F (Shared): number analyzed (Participants) | 833 | 280
  Serotype 7F (Shared) | 8.7 [8.1 to 9.3] | 10.1 [9.0 to 11.3]
  Serotype 9V (Shared): number analyzed (Participants) | 833 | 280
  Serotype 9V (Shared) | 7.6 [7.1 to 8.1] | 8.5 [7.6 to 9.5]
  Serotype 14 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 14 (Shared) | 10.3 [9.4 to 11.3] | 10.0 [8.5 to 11.8]
  Serotype 18C (Shared): number analyzed (Participants) | 833 | 280
  Serotype 18C (Shared) | 11.5 [10.7 to 12.4] | 9.3 [8.2 to 10.4]
  Serotype 19A (Shared): number analyzed (Participants) | 833 | 280
  Serotype 19A (Shared) | 6.4 [6.0 to 6.9] | 7.5 [6.7 to 8.5]
  Serotype 19F (Shared): number analyzed (Participants) | 833 | 280
  Serotype 19F (Shared) | 9.0 [8.3 to 9.7] | 9.8 [8.6 to 11.2]
  Serotype 23F (Shared): number analyzed (Participants) | 833 | 279
  Serotype 23F (Shared) | 10.8 [9.9 to 11.7] | 10.3 [9.0 to 11.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 833 | 280
  Serotype 22F (Unique to V114) | 8.9 [8.1 to 9.7] | 8.9 [7.5 to 10.7]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 833 | 280
  Serotype 33F (Unique to V114) | 6.4 [6.0 to 6.9] | 9.6 [8.4 to 11.1]

17. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Day 1 to Month 7
Description: as for outcome 11
Time Frame: Day 1 (Baseline) and Month 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 826 | 276
  Serotype 1 (Shared) | 87.7 [85.2 to 89.8] | 83.7 [78.8 to 87.9]
  Serotype 3 (Shared): number analyzed (Participants) | 820 | 270
  Serotype 3 (Shared) | 66.5 [63.1 to 69.7] | 66.7 [60.7 to 72.3]
  Serotype 4 (Shared): number analyzed (Participants) | 820 | 273
  Serotype 4 (Shared) | 84.3 [81.6 to 86.7] | 86.4 [81.8 to 90.3]
  Serotype 5 (Shared): number analyzed (Participants) | 831 | 279
  Serotype 5 (Shared) | 86.8 [84.3 to 89.0] | 87.1 [82.6 to 90.8]
  Serotype 6A (Shared): number analyzed (Participants) | 754 | 247
  Serotype 6A (Shared) | 73.5 [70.2 to 76.6] | 80.2 [74.6 to 84.9]
  Serotype 6B (Shared): number analyzed (Participants) | 802 | 273
  Serotype 6B (Shared) | 75.8 [72.7 to 78.7] | 74.4 [68.7 to 79.4]
  Serotype 7F (Shared): number analyzed (Participants) | 777 | 264
  Serotype 7F (Shared) | 59.8 [56.3 to 63.3] | 60.2 [54.0 to 66.2]
  Serotype 9V (Shared): number analyzed (Participants) | 810 | 273
  Serotype 9V (Shared) | 50.5 [47.0 to 54.0] | 52.4 [46.3 to 58.4]
  Serotype 14 (Shared): number analyzed (Participants) | 809 | 275
  Serotype 14 (Shared) | 64.9 [61.5 to 68.2] | 58.9 [52.8 to 64.8]
  Serotype 18C (Shared): number analyzed (Participants) | 805 | 273
  Serotype 18C (Shared) | 77.5 [74.5 to 80.4] | 76.2 [70.7 to 81.1]
  Serotype 19A (Shared): number analyzed (Participants) | 806 | 271
  Serotype 19A (Shared) | 68.2 [64.9 to 71.4] | 70.5 [64.7 to 75.8]
  Serotype 19F (Shared): number analyzed (Participants) | 818 | 272
  Serotype 19F (Shared) | 61.0 [57.6 to 64.4] | 62.9 [56.8 to 68.6]
  Serotype 23F (Shared): number analyzed (Participants) | 780 | 260
  Serotype 23F (Shared) | 73.5 [70.2 to 76.5] | 71.9 [66.0 to 77.3]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 742 | 254
  Serotype 22F (Unique to V114) | 59.0 [55.4 to 62.6] | 65.4 [59.2 to 71.2]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 810 | 273
  Serotype 33F (Unique to V114) | 53.3 [49.8 to 56.8] | 60.8 [54.7 to 66.6]

18. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Day 1 to Month 7
Description: as for outcome 12
Time Frame: Day 1 (Baseline) and Month 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 1 (Shared) | 81.4 [78.6 to 84.0] | 83.6 [78.7 to 87.7]
  Serotype 3 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 3 (Shared) | 40.7 [37.3 to 44.1] | 46.1 [40.1 to 52.1]
  Serotype 4 (Shared): number analyzed (Participants) | 830 | 278
  Serotype 4 (Shared) | 71.2 [68.0 to 74.3] | 82.0 [77.0 to 86.3]
  Serotype 5 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 5 (Shared) | 48.7 [45.3 to 52.2] | 51.8 [45.8 to 57.8]
  Serotype 6A (Shared): number analyzed (Participants) | 832 | 280
  Serotype 6A (Shared) | 81.6 [78.8 to 84.2] | 81.8 [76.8 to 86.1]
  Serotype 6B (Shared): number analyzed (Participants) | 832 | 280
  Serotype 6B (Shared) | 86.4 [83.9 to 88.7] | 85.4 [80.7 to 89.3]
  Serotype 7F (Shared): number analyzed (Participants) | 833 | 280
  Serotype 7F (Shared) | 77.4 [74.4 to 80.2] | 84.3 [79.5 to 88.3]
  Serotype 9V (Shared): number analyzed (Participants) | 833 | 280
  Serotype 9V (Shared) | 71.8 [68.6 to 74.8] | 77.1 [71.8 to 81.9]
  Serotype 14 (Shared): number analyzed (Participants) | 833 | 280
  Serotype 14 (Shared) | 76.7 [73.7 to 79.5] | 70.7 [65.0 to 76.0]
  Serotype 18C (Shared): number analyzed (Participants) | 833 | 280
  Serotype 18C (Shared) | 82.7 [80.0 to 85.2] | 80.4 [75.2 to 84.8]
  Serotype 19A (Shared): number analyzed (Participants) | 833 | 280
  Serotype 19A (Shared) | 65.8 [62.5 to 69.0] | 74.6 [69.1 to 79.6]
  Serotype 19F (Shared): number analyzed (Participants) | 833 | 280
  Serotype 19F (Shared) | 74.5 [71.4 to 77.5] | 78.9 [73.7 to 83.6]
  Serotype 23F (Shared): number analyzed (Participants) | 833 | 279
  Serotype 23F (Shared) | 77.8 [74.8 to 80.6] | 78.1 [72.8 to 82.8]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 833 | 280
  Serotype 22F (Unique to V114) | 68.8 [65.5 to 71.9] | 65.7 [59.8 to 71.3]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 833 | 280
  Serotype 33F (Unique to V114) | 68.2 [64.9 to 71.3] | 75.7 [70.3 to 80.6]

19. Secondary Outcome: GMFR in Serotype-specific OPA Month 6 to Month 7
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using the Multiplexed Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Month 6 (Baseline before Vaccination 2) and Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 839 | 280
  Serotype 1 (Shared) | 3.2 [2.9 to 3.5] | 2.0 [1.7 to 2.2]
  Serotype 3 (Shared): number analyzed (Participants) | 826 | 274
  Serotype 3 (Shared) | 2.0 [1.9 to 2.1] | 2.4 [2.2 to 2.7]
  Serotype 4 (Shared): number analyzed (Participants) | 837 | 281
  Serotype 4 (Shared) | 2.7 [2.5 to 2.9] | 1.7 [1.5 to 1.9]
  Serotype 5 (Shared): number analyzed (Participants) | 840 | 282
  Serotype 5 (Shared) | 2.7 [2.5 to 2.9] | 2.1 [1.9 to 2.4]
  Serotype 6A (Shared): number analyzed (Participants) | 818 | 270
  Serotype 6A (Shared) | 1.0 [1.0 to 1.1] | 1.1 [1.0 to 1.2]
  Serotype 6B (Shared): number analyzed (Participants) | 842 | 280
  Serotype 6B (Shared) | 1.1 [1.1 to 1.2] | 1.2 [1.1 to 1.4]
  Serotype 7F (Shared): number analyzed (Participants) | 837 | 281
  Serotype 7F (Shared) | 1.9 [1.8 to 2.0] | 1.4 [1.3 to 1.6]
  Serotype 9V (Shared): number analyzed (Participants) | 835 | 278
  Serotype 9V (Shared) | 1.6 [1.5 to 1.7] | 1.5 [1.4 to 1.7]
  Serotype 14 (Shared): number analyzed (Participants) | 841 | 280
  Serotype 14 (Shared) | 2.0 [1.8 to 2.1] | 1.5 [1.3 to 1.6]
  Serotype 18C (Shared): number analyzed (Participants) | 839 | 279
  Serotype 18C (Shared) | 1.3 [1.3 to 1.4] | 1.6 [1.4 to 1.7]
  Serotype 19A (Shared): number analyzed (Participants) | 830 | 282
  Serotype 19A (Shared) | 1.7 [1.6 to 1.8] | 1.5 [1.4 to 1.7]
  Serotype 19F (Shared): number analyzed (Participants) | 843 | 280
  Serotype 19F (Shared) | 1.9 [1.8 to 2.0] | 1.6 [1.5 to 1.8]
  Serotype 23F (Shared): number analyzed (Participants) | 837 | 280
  Serotype 23F (Shared) | 1.3 [1.2 to 1.4] | 1.4 [1.2 to 1.6]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 822 | 253
  Serotype 22F (Unique to V114) | 1.8 [1.7 to 1.9] | 9.6 [7.1 to 13.0]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 834 | 278
  Serotype 33F (Unique to V114) | 1.6 [1.5 to 1.8] | 6.5 [5.5 to 7.6]

20. Secondary Outcome: GMFR in Serotype-specific IgG Month 6 to Month 7
Description: IgG for the serotypes contained in Prevnar 13™ and V114 and (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. GMFR is the geometric mean of fold rise from baseline to postvaccination.
Time Frame: Month 6 (Baseline before Vaccination 2) and Month 7
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 1 (Shared) | 2.1 [2.0 to 2.2] | 1.5 [1.4 to 1.7]
  Serotype 3 (Shared): number analyzed (Participants) | 842 | 282
  Serotype 3 (Shared) | 1.7 [1.6 to 1.7] | 2.0 [1.8 to 2.1]
  Serotype 4 (Shared): number analyzed (Participants) | 840 | 280
  Serotype 4 (Shared) | 2.0 [1.9 to 2.1] | 1.6 [1.5 to 1.7]
  Serotype 5 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 5 (Shared) | 1.9 [1.8 to 1.9] | 1.5 [1.4 to 1.6]
  Serotype 6A (Shared): number analyzed (Participants) | 842 | 282
  Serotype 6A (Shared) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1]
  Serotype 6B (Shared): number analyzed (Participants) | 843 | 282
  Serotype 6B (Shared) | 1.1 [1.0 to 1.1] | 1.2 [1.2 to 1.3]
  Serotype 7F (Shared): number analyzed (Participants) | 843 | 282
  Serotype 7F (Shared) | 1.7 [1.6 to 1.8] | 1.4 [1.3 to 1.5]
  Serotype 9V (Shared): number analyzed (Participants) | 841 | 282
  Serotype 9V (Shared) | 1.5 [1.5 to 1.6] | 1.4 [1.3 to 1.5]
  Serotype 14 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 14 (Shared) | 1.7 [1.6 to 1.8] | 1.4 [1.3 to 1.5]
  Serotype 18C (Shared): number analyzed (Participants) | 843 | 282
  Serotype 18C (Shared) | 1.1 [1.0 to 1.1] | 1.1 [1.1 to 1.2]
  Serotype 19A (Shared): number analyzed (Participants) | 842 | 282
  Serotype 19A (Shared) | 1.4 [1.3 to 1.4] | 1.4 [1.3 to 1.4]
  Serotype 19F (Shared): number analyzed (Participants) | 843 | 282
  Serotype 19F (Shared) | 1.6 [1.6 to 1.7] | 1.6 [1.5 to 1.7]
  Serotype 23F (Shared): number analyzed (Participants) | 842 | 281
  Serotype 23F (Shared) | 1.1 [1.1 to 1.2] | 1.2 [1.1 to 1.2]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 843 | 282
  Serotype 22F (Unique to V114) | 1.8 [1.7 to 1.9] | 8.8 [7.4 to 10.4]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 843 | 282
  Serotype 33F (Unique to V114) | 1.6 [1.6 to 1.7] | 9.9 [8.6 to 11.3]

21. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Month 6 to Month 7
Description: as for outcome 11
Time Frame: Month 6 (Baseline before Vaccination 2) and Month 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 839 | 280
  Serotype 1 (Shared) | 40.2 [36.8 to 43.6] | 21.4 [16.8 to 26.7]
  Serotype 3 (Shared): number analyzed (Participants) | 826 | 274
  Serotype 3 (Shared) | 19.2 [16.6 to 22.1] | 25.5 [20.5 to 31.1]
  Serotype 4 (Shared): number analyzed (Participants) | 837 | 281
  Serotype 4 (Shared) | 30.8 [27.7 to 34.1] | 14.9 [11.0 to 19.7]
  Serotype 5 (Shared): number analyzed (Participants) | 840 | 282
  Serotype 5 (Shared) | 32.5 [29.3 to 35.8] | 23.0 [18.3 to 28.4]
  Serotype 6A (Shared): number analyzed (Participants) | 818 | 270
  Serotype 6A (Shared) | 3.9 [2.7 to 5.5] | 5.9 [3.4 to 9.4]
  Serotype 6B (Shared): number analyzed (Participants) | 842 | 280
  Serotype 6B (Shared) | 4.6 [3.3 to 6.3] | 6.4 [3.9 to 10.0]
  Serotype 7F (Shared): number analyzed (Participants) | 837 | 281
  Serotype 7F (Shared) | 14.6 [12.3 to 17.2] | 7.5 [4.7 to 11.2]
  Serotype 9V (Shared): number analyzed (Participants) | 835 | 278
  Serotype 9V (Shared) | 11.9 [9.7 to 14.2] | 10.4 [7.1 to 14.6]
  Serotype 14 (Shared): number analyzed (Participants) | 841 | 280
  Serotype 14 (Shared) | 17.8 [15.3 to 20.6] | 8.6 [5.6 to 12.5]
  Serotype 18C (Shared): number analyzed (Participants) | 839 | 279
  Serotype 18C (Shared) | 5.4 [3.9 to 7.1] | 14.3 [10.4 to 19.0]
  Serotype 19A (Shared): number analyzed (Participants) | 830 | 282
  Serotype 19A (Shared) | 15.9 [13.5 to 18.6] | 12.1 [8.5 to 16.4]
  Serotype 19F (Shared): number analyzed (Participants) | 843 | 280
  Serotype 19F (Shared) | 17.7 [15.2 to 20.4] | 12.9 [9.2 to 17.4]
  Serotype 23F (Shared): number analyzed (Participants) | 837 | 280
  Serotype 23F (Shared) | 9.2 [7.3 to 11.4] | 11.4 [7.9 to 15.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 822 | 253
  Serotype 22F (Unique to V114) | 16.7 [14.2 to 19.4] | 52.6 [46.2 to 58.9]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 834 | 278
  Serotype 33F (Unique to V114) | 15.8 [13.4 to 18.5] | 62.6 [56.6 to 68.3]

22. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Month 6 to Month 7
Description: as for outcome 12
Time Frame: Month 6 (Baseline before Vaccination 2) and Month 7
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 1133 | 379
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 1 (Shared) | 16.4 [13.9 to 19.0] | 8.2 [5.2 to 12.0]
  Serotype 3 (Shared): number analyzed (Participants) | 842 | 282
  Serotype 3 (Shared) | 6.3 [4.8 to 8.2] | 13.8 [10.0 to 18.4]
  Serotype 4 (Shared): number analyzed (Participants) | 840 | 280
  Serotype 4 (Shared) | 15.2 [12.9 to 17.8] | 7.5 [4.7 to 11.2]
  Serotype 5 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 5 (Shared) | 12.1 [10.0 to 14.5] | 5.7 [3.3 to 9.1]
  Serotype 6A (Shared): number analyzed (Participants) | 842 | 282
  Serotype 6A (Shared) | 0.6 [0.2 to 1.4] | 1.1 [0.2 to 3.1]
  Serotype 6B (Shared): number analyzed (Participants) | 843 | 282
  Serotype 6B (Shared) | 0.7 [0.3 to 1.5] | 2.8 [1.2 to 5.5]
  Serotype 7F (Shared): number analyzed (Participants) | 843 | 282
  Serotype 7F (Shared) | 8.4 [6.6 to 10.5] | 4.3 [2.2 to 7.3]
  Serotype 9V (Shared): number analyzed (Participants) | 841 | 282
  Serotype 9V (Shared) | 6.3 [4.8 to 8.2] | 3.9 [2.0 to 6.9]
  Serotype 14 (Shared): number analyzed (Participants) | 843 | 282
  Serotype 14 (Shared) | 9.8 [7.9 to 12.1] | 3.9 [2.0 to 6.9]
  Serotype 18C (Shared): number analyzed (Participants) | 843 | 282
  Serotype 18C (Shared) | 0.6 [0.2 to 1.4] | 0.7 [0.1 to 2.5]
  Serotype 19A (Shared): number analyzed (Participants) | 842 | 282
  Serotype 19A (Shared) | 3.4 [2.3 to 4.9] | 4.3 [2.2 to 7.3]
  Serotype 19F (Shared): number analyzed (Participants) | 843 | 282
  Serotype 19F (Shared) | 8.1 [6.3 to 10.1] | 6.4 [3.8 to 9.9]
  Serotype 23F (Shared): number analyzed (Participants) | 842 | 281
  Serotype 23F (Shared) | 0.5 [0.1 to 1.2] | 1.1 [0.2 to 3.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 843 | 282
  Serotype 22F (Unique to V114) | 10.2 [8.2 to 12.4] | 64.9 [59.0 to 70.5]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 843 | 282
  Serotype 33F (Unique to V114) | 7.5 [5.8 to 9.5] | 75.9 [70.5 to 80.8]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after each vaccination; Serious adverse events and all-cause mortality: Up to Month 7 (Up to 44 days after vaccination 2).
Description: The analysis population included all randomized participants who received the relevant study vaccination for the timepoint of interest and were included in the intervention group according to the intervention they received. One participant in the Prevnar 13™ group incorrectly received V114 and was included in the V114 group for safety analyses.
Groups:
- V114 (Post-PNEUMOVAX™23): Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
- Prevnar 13™ (Post-PNEUMOVAX™23): Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Month 6 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™ | V114 (Post-PNEUMOVAX™23) | Prevnar 13™ (Post-PNEUMOVAX™23)
All-Cause Mortality (participants affected / at risk) | 4/1134 | 2/378 | 0/1036 | 0/345
Serious Adverse Events (participants affected / at risk) | 49/1134 | 12/378 | 3/1036 | 3/345
Other Adverse Events (participants affected / at risk) | 934/1134 | 298/378 | 771/1036 | 258/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=1134) | Prevnar 13™ (N=378) | V114 (Post-PNEUMOVAX™23) (N=1036) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=345)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Physical assault (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=1134) | Prevnar 13™ (N=378) | V114 (Post-PNEUMOVAX™23) (N=1036) | Prevnar 13™ (Post-PNEUMOVAX™23) (N=345)
Fatigue (General disorders) | 389 (510) | 139 (186) | 312 (366) | 106 (139)
Injection site erythema (General disorders) | 174 (180) | 56 (57) | 235 (237) | 88 (91)
Injection site pain (General disorders) | 865 (931) | 260 (292) | 714 (762) | 231 (252)
Injection site swelling (General disorders) | 251 (257) | 84 (84) | 305 (307) | 113 (113)
Arthralgia (Musculoskeletal and connective tissue disorders) | 144 (180) | 44 (63) | 124 (130) | 38 (47)
Myalgia (Musculoskeletal and connective tissue disorders) | 327 (377) | 100 (113) | 250 (260) | 88 (99)
Headache (Nervous system disorders) | 300 (425) | 94 (122) | 220 (274) | 73 (93)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03547167/Prot_SAP_000.pdf